CLINICAL TRIAL: NCT00152698
Title: A Randomised, Double-blind, Placebo-controlled, Phase III Trial to Study the Effect of Irbesartan on Endothelial Function of the Retinal Vasculature in Patients With Hypercholesterolemia
Brief Title: Effect of Irbesartan on Endothelial Function of the Retinal Vasculature in Patients With Hypercholesterolemia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never active
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Roland E. Schmieder, Prof. Dr. med., University of Erlangen-Nürnberg Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Retina-Irbesartan
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irbesartan (Active Comparator)
  Interventions: Drug: Irbesartan
- Placebo (Placebo Comparator)
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan

SUMMARY:
The retinal vasculature is morphologically and functionally related to the cerebral vessels due to its common origin from the internal carotid artery. A recent study demonstrated that endothelium-dependent vasodilation of the retinal vasculature is impaired in patients with essential hypertension, which is a strong risk factor for stroke. Furthermore, AT1-receptor blockade was demonstrated to improve retinal endothelium-dependent vasodilation in these hypertensive patients. Hypercholesterolemia is also a risk factor for ischemic stroke and impairment of endothelial function has been observed in various vascular beds in hypercholesterolemic patients, including the coronary and the forearm vasculature. Whether endothelial function of the retinal vasculature is impaired in patients with hypercholesterolemia has not yet been investigated. In patients with stroke, AT1-receptor blockade and angiotensin-converting enzyme inhibition have beneficial effects on clinical outcome. Alterations of endothelial function of the cerebral vasculature might be one pathogenetic factor for the beneficial clinical outcome. To further address this issue, the present study was designed to test the hypothesis that endothelium-dependent vasodilation of the retinal vasculature is impaired in hypercholesterolemic patients and that endothelial function can be improved by AT1-receptor blockade.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18-65 years with LDL-cholesterol >= 130mg/dl
* Male healthy control subjects aged 18-65 years

Exclusion Criteria:

* All kinds of secondary hyperlipidemia.
* Advanced damage of vital organs (grades III and IV retinopathy)
* Lipid-lowering drugs (including lipid lowering dietary supplements or food additives) within the last 4 weeks
* History of serious hypersensitivity reaction to AT1-receptor blockers
* Actual or anamnestic alcohol- or drug abuse.
* Smokers or ex-smokers < 1 year.
* Patients with Diabetes mellitus (oral medication or insulin).
* Patients with arterial fibrillation or AV-Block (II° or more).
* Patients with anamnestic myocardial infarction.
* Patients with instable angina pectoris including EcG-aberrations or cardiac insufficiency NYHA III or IV.
* History of malignancy (unless a documented disease-free period exceeding 10 years is present) with the exception of basal cell carcinoma of the skin
* History of allograft transplantation
* Patients with anaphylaxis or known therapy resistance of the used test matters
* Therapy with not approved concomitant medication, or participation in a clinical study within 4 weeks preceding treatment start.
* Disease which interfere with the pharmacodynamics and pharmacokinetics of the study drug.
* Liver or kidney disease with SGOT, GPT, g-GT, AP, bilirubin and creatinin above 200% of standard.
* Patients, who are not sufficiently compliant, or patients, who are not capable or willing to appear for controlling visits.
* Presumed risk of transmission of HIV or hepatitis via blood from the proband

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11 (Estimated); Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of retinal endothelial function between hypercholesterolemic patients and healthy control subjects

SECONDARY OUTCOMES:
Effect of AT1-receptor blockade on retinal endothelial function in hypercholesterolemic patients

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, MD, Principal Investigator — CRC, Medizinische Klinik 4, Nephrology and Hypertension, University of Erlangen-Nürnberg
Locations (1):
- CRC, Medizinsiche Klinik 4, Nephrology and Hypertension, University of Erlangen-Nürnberg, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Kannenkeril D, Bosch A, Harazny J, Karg M, Jung S, Ott C, Schmieder RE. Early vascular parameters in the micro- and macrocirculation in type 2 diabetes. Cardiovasc Diabetol. 2018 Sep 19;17(1):128. doi: 10.1186/s12933-018-0770-4. PMID 30231923
- [Derived] Bosch AJ, Harazny JM, Kistner I, Friedrich S, Wojtkiewicz J, Schmieder RE. Retinal capillary rarefaction in patients with untreated mild-moderate hypertension. BMC Cardiovasc Disord. 2017 Dec 21;17(1):300. doi: 10.1186/s12872-017-0732-x. PMID 29268712
- [Derived] Jumar A, Harazny JM, Ott C, Kistner I, Friedrich S, Schmieder RE. Improvement in Retinal Capillary Rarefaction After Valsartan Treatment in Hypertensive Patients. J Clin Hypertens (Greenwich). 2016 Nov;18(11):1112-1118. doi: 10.1111/jch.12851. Epub 2016 Jun 16. PMID 27306560